CLINICAL TRIAL: NCT04376060
Title: The Horizontal Ridge Augmentation Using Equine Xenograft and a Collagenated Porcine Cortical Lamina: A Clinical, Radiographic and Histological Prospective Study
Brief Title: The Horizontal Ridge Augmentation Using Equine Xenograft and a Collagenated Porcine Cortical Lamina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Sarah Khalil, Principal Investigator, Saint-Joseph University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMD 141
Record Dates: First submitted 2020-04-28; First posted 2020-05-06 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Horizontal Ridge Deficiency
Keywords: osteogenesis; xenograft; membrane

STUDY DESIGN:
Intervention Model Description: Fourteen patients (1 male, 13 females) aged between 27 and 64 years old were selected from the Department of Periodontology of the Faculty of Dentistry, Saint Joseph University Beirut.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study population (Experimental): Fifteen patients (1 male, 14 females) aged between 27 and 64 years old
  Interventions: Device: Gen-Os®; The soft lamina (OsteoBiol®)

INTERVENTIONS:
Device: Gen-Os®; The soft lamina (OsteoBiol®) — The xenograft used in this study was the Gen-Os® by OsteoBiol; as described by the manufacturer, it is a carbonated nanocrystal bone mineral and collagen of natural heterologous origin, obtained by the treatment of cortical bone tissue of equine origins. Its granulometry ranges between 0.25 to 1 mm and it is described as being slightly radiopaque.
  The soft lamina (OsteoBiol®) used is a 35x35mm medium curved membrane of porcine origins. Its clinical indications as described by the fabricator: a co-adjuvant for the reconstruction or the partial or complete recovery of lost bone portions, fillers of non-infected, non-sclerotic and well blood bedewed bone defects.

SUMMARY:
The primary aim of this study is to clinically, radiographically and histologically evaluate the lateral bone augmentation of the soft porcine cortical lamina (OsteoBiol®) using equine-derived bone particles (OsteoBiol®)

DETAILED DESCRIPTION:
The xenograft used in this study was the Gen-Os® by OsteoBiol; The soft lamina (OsteoBiol®) used is a 35x35mm medium curved membrane of porcine origins.

The fixation system used was the Pro-fix™ Precision Fixation System, consisting of self-drilling membrane fixation screws of 1.5 mm x 3.0 mm.

Fifteen patients (1 male, 14 females) aged between 27 and 64 years old were selected from the Department of Periodontology of the Faculty of Dentistry, Saint Joseph University Beirut.

Clinical and radiographic examinations were done prior to any procedure. The edentulous area was examined to identify the availability of keratinised mucosa and the possibility of implant placement in the mesio-distal and inter-arch planes. Radiographic examination was completed using a cone beam computed tomography (CBCT) scan of the affected region, where the indication for vertical augmentation was selected and excluded from the study. All the patients were given oral hygiene instructions and prophylaxis.

Each patient received 2g of Amoxicillin one hour prior to surgery. Patients were instructed to mouthrinse with chlorhexidine 0.12% gluconate mouthwash for 1 minute. Extra-oral disinfection was made using topical chlorhexidine.

Local and/or regional anaesthesia was obtained using Septanest® (Articaine hydrochloride 4% with adrenaline 1:100,000) A mid-crestal incision was performed and extended into the sulcus of the adjacent teeth, if present. At least one vertical releasing incision extending beyond the muco-gingival junction was made. A muco-periosteal flap of full thickness was raised and extended buccally, whereas palatally it was reflected to expose 3 mm of bone. Lingually the flap was elevated until reaching the mylo-hyoid line. Decortication was carried out using a twist drill with a stop of 3mm of length to ensure a good perfusion of the graft.

The soft cortical lamina had been soaked in saline sterile water since the beginning of the surgery in order to achieve good elasticity and easier manipulation. It was then trimmed with sterile scissors and adapted to the recipient site while making sure it was not in contact with the surrounding teeth. It was first fixed on the palatal/lingual side. The cortico-cancellous heterologous bone mix which was previously hydrated in sterile saline for ten minutes, was placed on the ridge in sufficient quantities and covered by the membrane while being adapted in the desired shape of the future ridge. The membrane was reclined and also fixated on the buccal side for better adaptability and immobilization. In order to ensure a tension free closure, the buccal flap was advanced using a periosteal releasing incision connecting the vertical incisions thus achieving elasticity of the flap. Precaution was taken to identify and carefully isolate the mental nerve from the surrounding tissues when present. The lingual flaps were advanced using a blunt instrument to detach the muscular insertion of the mylo-hyoid from the lingual flap.

Once proper elasticity was achieved, horizontal mattress sutures were placed at 4mm from the incision line using a non-resorbable polytetrafluroethylene (PTFE) 4/0 monofilament suture.

They were followed by single interrupted sutures close to the edges of the flap in order to create a connective tissue-connective tissue contact, thus creating a barrier to reduce the incidence of membrane exposure.

All patients were instructed to receive an injection of betamethasone dipropionate and disodium phosphate directly after the surgery and received 2g of Amoxicillin per day for a total of 7 days.

Post-operative recommendations were clearly written and given to the patient. Chlorhexidine was prescribed starting the second day after surgery until suture removal.

Sutures were removed at 14 days, they were left for another 7 days when found necessary to secure the healing.

At 6 months from the surgery, a CBCT scan of the grafted area was taken and measures were made for the choice of the implant diameter and length. In all of the post-operative CBCTs, implant placement seemed possible.

On the day of the implant placement, local anaesthesia was made, followed by a mid-crestal incision and occasionally a vertical one, allowing access to the fixation screws for their removal.

A biopsy was taken at the site of implant placement using a trephine burr of outer diameter of 3.5mm and inner diameter of 2.5mm. The trephine and bone were immersed in 10% buffered formaldehyde and fixated for histology. The implants (Straumann®, Bone Level Cylindrical) were placed at the corresponding sites of the biopsies, and the choice of a cover or a healing screw was made depending on the clinical situation and the primary stability of the implant.

Implant insertion torques were noted as indicated on the implant torque wrench. Periapical radio-graphs were taken, the flap was sutured and the patients received a daily dose of 2g of Amoxicillin for 7 days and diclofenac potassium inflammatory for pain management. They were also notified to mouth rinse with Chlorhexidine 0.12% for 10 days.

Radiological protocol

Image acquisition:

At consultation and six months after the regeneration procedure, patients were scanned with the Newton VGI CBCT machine. Imaging conditions were: 110 kv tube voltage; 2.2 to 8.30 milliampere (mA) tube current; 15 x 15 cm field of view; and 0.3 mm voxel size. Projection data were collected with a device rotating 360 degrees around patients over a total acquisition time of 18 seconds.

Evaluation of images:

Scan data were saved in DICOM (Digital Imaging and Communications in Medicine) format and image analysis and measurements were performed using the Blue Sky Plan® (Blue Sky Bio, LLC, Grayslake, IL, USA) which provided axial, coronal and sagittal views through multiplanar reconstructions of 0.3 mm slices. Axial images were reoriented to occlusal plane when present or to palatal plane as a horizontal reference. A panoramic curve was created and cross-sectional images perpendicular to that curve were reconstructed at a 1 mm interval.

Advanced jaw segmentation:

For each scan, an advanced jaw segmentation technique was realized using the Blue Sky Plan software by means of threshold segmentation and contour interpolation. First the region of interest (corresponding jaw) was selected on the panoramic view. Second, several axial, coronal and cross-sectional slices equally distributed/chosen by the software were used to draw the outline of the bone. This created a matrix to the final automatic segmentation step by the software to finalize the segmentation data and create a 3D model of the jaw. Finally, the outline of the 3D model was checked and adjusted manually on the 2D slices in all the planes in cases of over or missing contour. The result was an accurate 3D model of the corresponding jaw.

Virtual implant placement and jaw superimposition:

On the post-operative CBCT plan, virtual implants were placed in the optimal position regarding bone and prosthetic reference when present.

In order to compare directly the pre and post-operative models, the pre-operative bone model was loaded into the post-operative plan an n-point registration technique was used for the superimposition of the two models. The outline of each model was visible in a unique color for comparison.

A vestibulo-lingual implant centric section perpendicular to the panoramic curve and parallel to the long axis of the simulated implant was used to make all the measurements as follow:

Horizontal bone width measurements

For each implant site, pre and post-operative horizontal bone width were measured at 4 levels. Bone width was calculated from the distance between the most buccal and most lingual bone points at each level while being parallel to the simulated implant platform.

* H0-T1 and H0-T2: Pre and post-operative horizontal bone width at implant platform level.
* H2-T1 and H2-T2: Pre and post-operative horizontal bone width at 2mm apically to implant platform.
* H4-T1 and H4-T2: Pre and post-operative horizontal bone width at 4mm apically to implant platform.

Vertical bone gain/loss measurements

For each implant site, pre and post-operative vertical bone gain were measured at 3 levels. Vertical bone gain/loss was calculated from the distance between the most coronal pre-operative bone points.

Histology

Fixation and inclusion:

Samples were taken at six months after regeneration and were treated with non-demineralized histology. They were fixed in LILLIE neutral formalin, diluted to 10% in buffered sodium phosphate pH 7.4. The fixation period lasted 3 weeks. The samples were then rinsed under running water for 48 hours.

The dehydration of the samples was carried out in alcohol baths of increasing concentrations for 48 hours, then the clarification, allowing the penetration of methacrylate, in 2 successive xylene baths of 24 hours each.

Cutting technique:

The blocks were cut under irrigation and at slow speed with an Exact saw (Cutting machine EXACT-APPARATEBAU Nordersted, Germany), so as to take cuts of at least 80 μm. These cuts were subsequently reduced in thickness with the Exact abrasion system. The polishing was carried out with abrasive paper discs of decreasing granulometry making it possible to reduce the thickness of the cuts automatically to the desired value. The cuts were separated into S (superficial), M (median) and P (profound) cuts, the superficial ones being the cuts facing the periosteum.

Staining:

The sections were stained with Giemsa-Paragon and basic fuchsin. Giemsa will give cells and nuclei the color blue, and Paragon will stain bone in red.

Histomorphometry:

The qualitative observation of the sections was done under a digital microscope (Keyence digital microscope VHX-6000) with normal and polarized light visualisations. For histological quantification, an optical microscope was used (Olympus BX 60, Olympus Corporation, Tokyo, Japan) connected to a digital camera (Olympus E330), along with the software Image J/ Fiji.

It was first calibrated by measuring the scale bar present on the image. The image was made into black and white (Type: 8-bit). The scale was set by measuring the length of the scale bar in pixels and by setting its known distance in millimetres. It was then set as 'Global' for all the images with the same scale.

The total area of the concerned section was measured. Then the bone and osteoid volume were quantified using the Bone Volume Mask and by using the 'wand tool' to select all the black areas. The percentage of bone and osteoid matrix in each section was consequently calculated.

Statistical analysis:

The statistical package software for social sciences (SPSS for Windows, Chicago, IL, USA, version 25.0) was performed for statistical analysis of the data. The alpha error was set at -p-value<0.05. Frequency and percentage were utilized to describe categorical variables. Mean and standard-deviation were used for continuous variables.

* Repeated measure analysis of variance with two within-subjects factors (Time: Baseline and six months; distance: 0mm, 2mm, 4mm, and 6 mm) was performed to compare the mean bone level within groups. It was followed by univariate analyses and Bonferroni post hoc tests.
* Repeated measure analysis of variance with one within-subjects factor (distance: 0mm, 2mm, 4mm, and 6 mm) followed by Bonferroni post hoc tests was used to compare the mean horizontal gain.
* Repeated measure analysis of variance with one within-subjects factor (level: buccal, median, lingual) followed by Bonferroni post hoc tests was executed to compare the mean vertical gain.
* One sample t tests were used to compare the mean vertical gain with a theoretical value "0'' that supposed the absence of gain.
* Student t tests were performed to compare continuous variables between two groups.
* Pearson correlation coefficients were calculated to assess the relationship between continuous variables.
* Kruskal-Wallis tests were used to compare histomorphometric measurements between different levels.

ELIGIBILITY:
Inclusion Criteria:

* systematically healthy
* good oral hygiene (FMPS and FMBS <20%).
* having ridges with deficiencies in width (<4 mm, Cawood and Howell class IV) which did not allow correct implant placement.

Exclusion Criteria:

* pregnant and lactating women,
* patients suffering from a systematic disease
* patients on bisphosphonates
* smokers (>10 cigarettes/day)
* patients needing vertical augmentations

Ages: 27 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Chakar, PhD, Study Director — Saint-Joseph University
Locations (1):
- Sarah Khalil, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As soon as the study is published (summer 2020)
Access Criteria: Publication in a scientific journal

REFERENCES:
- [Background] Rossi R, Rancitelli D, Poli PP, Rasia Dal Polo M, Nannmark U, Maiorana C. The use of a collagenated porcine cortical lamina in the reconstruction of alveolar ridge defects. A clinical and histological study. Minerva Stomatol. 2016 Oct;65(5):257-68. PMID 27580650
- [Background] Deepika-Penmetsa SL, Thomas R, Baron TK, Shah R, Mehta DS. Cortical lamina technique: A therapeutic approach for lateral ridge augmentation using guided bone regeneration. J Clin Exp Dent. 2017 Jan 1;9(1):e21-e26. doi: 10.4317/jced.53008. eCollection 2017 Jan. PMID 28149458
- [Background] Wachtel H, Fickl S, Hinze M, Bolz W, Thalmair T. The bone lamina technique: a novel approach for lateral ridge augmentation--a case series. Int J Periodontics Restorative Dent. 2013 Jul-Aug;33(4):491-7. doi: 10.11607/prd.1248. PMID 23820709

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: Patients who complied with the inclusion criteria of this study and received the procedure of horizontal bone augmentation.
Period: Overall Study
Arm/Group | Study Population
Started | 15
Completed | 14
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Population: Patients who received the intervention of horizontal bone augmentation using the cortical lamina and the equine-derived bone particles,
Arm/Group | Study Population
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Horizontal bone augmentation at 0 mm [Mean (Standard Deviation); unit: mm] — Measured in mm at the top of the crest at the regenration site
  mm | 2.989 (1.612)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Radiological Bone Width Augmentation at 0 mm
Description: Width difference measured at the top of the crest (0 mm) at the site of implant placement, measured in mm over superimposition of pre-operative (baseline) Cone Beam Computed Tomography and postoperative (at 6 months) Cone Beam Computed Tomography (CBCT).
  The value measured at 6 months minus the value measured at baseline = width difference measured at top of the crest (0 mm).
Time Frame: Six months after the regeneration procedure
Population: 14 patients who have had the regeneration procedure
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Study Population: Fourteen patients (1 male, 13 females) aged between 27 and 64 years old
Arm/Group | Study Population
Number analyzed (Participants) | 14
mm | 2.274 (1.517)

2. Primary Outcome: Change From Baseline in Radiological Bone Width Augmentation at 2 mm
Description: Width difference measured at 2 mm of the top of the crest at the site of implant placement, measured in mm over superimposition of pre-operative (baseline) Cone Beam Computed Tomography and postoperative (at 6 months) Cone Beam Computed Tomography (CBCT).
  The value measured at 6 months minus the value measured at baseline = width difference measured at 2 mm of the top of the crest.
Time Frame: Six months after the regeneration procedure
Population: 14 patients who have had the regeneration procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Study Population
Number analyzed (Participants) | 14
mm | 2.274 (1.015)

3. Primary Outcome: Change From Baseline in Radiological Bone Width Augmentation at 4 mm
Description: Width difference measured at 4 mm of the top of the crest at the site of implant placement, measured in mm over superimposition of pre-operative (baseline) Cone Beam Computed Tomography and postoperative (at 6 months) Cone Beam Computed Tomography (CBCT).
  The value measured at 6 months minus the value measured at baseline = width difference measured at 4 mm of the top of the crest.
Time Frame: Six months after the regeneration procedure
Population: 14 patients who have had the regeneration procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Study Population
Number analyzed (Participants) | 14
mm | 2.028 (0.79)

4. Primary Outcome: Change From Baseline in Radiological Bone Width Augmentation at 6 mm
Description: Width difference measured at 6 mm of the top of the crest at the site of implant placement, measured in mm over superimposition of pre-operative (baseline) Cone Beam Computed Tomography and postoperative (at 6 months) Cone Beam Computed Tomography (CBCT).
  The value measured at 6 months minus the value measured at baseline = width difference measured at 6 mm of the top of the crest.
Time Frame: Six months after the regeneration procedure
Population: 14 patients who have had the regeneration procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Study Population
Number analyzed (Participants) | 14
mm | 1.442 (0.929)

5. Secondary Outcome: Number of Implants Placed at 6 Months From the Regeneration Procedure
Description: Number of implants placed in the regenerated areas at 6 months from the regeneration procedure
Time Frame: Six months after the regeneration procedure
Measure: Number; unit: Implants
Arm/Group | Study Population
Number analyzed (Participants) | 14
Implants | 26

6. Secondary Outcome: Change From Baseline in Radiological Bone Height Augmentation in mm Measured Buccally
Description: Height difference measured buccally in mm at the site of implant placement, measured over superimposition of pre-operative Cone Beam Computed Tomography (baseline) and post-operative Cone Beam Computed Tomography (at 6 months) The value measured at 6 months minus the value measured at baseline = height difference measured buccally
Time Frame: Six months after the regeneration procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Study Population
Number analyzed (Participants) | 14
mm | 2.776 (2.445)

7. Secondary Outcome: Bone Percentage Superficially
Description: The percentage of bone in the superficial cuts
Time Frame: Six months after the regeneration procedure
Measure: Mean (Standard Deviation); unit: percentage of bone tissue
Arm/Group | Study Population
Number analyzed (Participants) | 14
percentage of bone tissue | 60.781 (11.629)

8. Secondary Outcome: Change From Baseline in Radiological Bone Height Augmentation in mm Measured Medially
Description: Height difference measured medially in mm at the site of implant placement, measured over superimposition of pre-operative Cone Beam Computed Tomography (baseline) and post-operative Cone Beam Computed Tomography (at 6 months) The value measured at 6 months minus the value measured at baseline = height difference measured medially
Time Frame: Six months after the regeneration procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Study Population
Number analyzed (Participants) | 14
mm | 0.812 (0.905)

9. Secondary Outcome: Change From Baseline in Radiological Bone Height Augmentation in mm Measured Lingually
Description: Height difference measured lingually in mm at the site of implant placement, measured over superimposition of pre-operative Cone Beam Computed Tomography (baseline) and post-operative Cone Beam Computed Tomography (at 6 months) The value measured at 6 months minus the value measured at baseline = height difference measured lingually
Time Frame: Six months after the regeneration procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Study Population
Number analyzed (Participants) | 14
mm | 0.734 (0.812)

10. Secondary Outcome: Bone Percentage Medially
Description: The percentage of bone in the median cuts
Time Frame: Six months after the regeneration procedure
Measure: Mean (Standard Deviation); unit: percentage of bone tissue
Arm/Group | Study Population
Number analyzed (Participants) | 14
percentage of bone tissue | 73.616 (14.136)

11. Secondary Outcome: Bone Percentage in the Deep Cuts
Description: The percentage of bone in the deep cuts
Time Frame: Six months after the regeneration procedure
Measure: Mean (Standard Deviation); unit: percentage of bone tissue
Arm/Group | Study Population
Number analyzed (Participants) | 14
percentage of bone tissue | 77.234 (7.183)

ADVERSE EVENTS:
Time Frame: 6 months
Description: The risk of Serious Adverse Events and All-Cause Mortality after Guided Bone Regeneration in healthy patients is null when the practitioner has made a thorough investigation of the medical history of the patient. This is not a life-threatening procedure
Arm/Group | Study Population
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Population (N=15)
Bone Regeneration Failure (Injury, poisoning and procedural complications) | 1 (1) — A complication of the bone regeneration procedure: the grafted bone was not successfully integrated. It was removed during the implant placement surgery, and no implants were placed.

LIMITATIONS AND CAVEATS:
Technical problems with histomorphometric measurements: the distinction between pre-existent and newly formed bone was not possible in all the histological cuts

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT04376060/ICF_000.pdf
  • Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT04376060/SAP_001.pdf
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT04376060/Prot_002.pdf